CLINICAL TRIAL: NCT04178161
Title: Image Guided Targeted Photoablation for the Treatment of Localized Hyperhidrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Sciton (Industry)
Responsible Party: Principal Investigator, Richard Rox Anderson, MD, Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016P001071
Record Dates: First submitted 2019-09-17; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis | interventions — Laser Therapy

STUDY DESIGN:
Intervention Model Description: The study involves a single group of patients with Hyperhidrosis. Left and right palms are randomized for treatment versus control (untreated).
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treated side (Experimental): Two regions are designated on the upper back. Randomized to treatment and control sides.
  Treatment side receives laser treatment of the sweat glands.
  Interventions: Device: Laser treatment
- Untreated side (No Intervention): Two regions are designated on the upper back. Randomized to treatment and control sides.
  Control side is untreated.

INTERVENTIONS:
Device: Laser treatment — Iontophoresis of methylene blue is used to identify the sweat glands. An image guided fractional erbium laser is used to specifically target these glands for ablation.
  Arms: Treated side

SUMMARY:
Hyperhidrosis is a condition in which sweating is in excess of that required for normal regulation of body temperature. Commonly affected areas in primary hyperhidrosis include axillae, palms and soles. Secondary hyperhidrosis can affect scalp, face, neck, back, groin and legs. Hyperhidrosis can negatively impact, employment, relationships, or other aspects of quality of life.

The investigators propose to investigate the use of a unique image-guided laser to specifically ablate eccrine sweat glands.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of ages between 18 and 65 years.
2. Subjects with any Fitzpatrick skin type.
3. Subjects who are proficient in the English language.
4. Willingness to participate in the study.
5. Willingness to undergo experimental procedure.
6. Informed consent agreement signed by the subject.
7. Willingness to follow the follow-up schedule.
8. Willingness not to use any other hyperhidrosis treatment to the tests sites during the study period (i.e. deodorant, at-home iontophoresis, Botox, MiraDry).
9. Patient rates symptoms at level "3" or "4" on the hyperhidrosis disease severity scale (HDSS, see below).
10. Subject in appropriate physical health to ride a stationary bicycle to the point of eliciting sweat.
11. No known allergy to iodine or potato starch

Exclusion Criteria:

1. Pregnancy
2. Subjects on systemic treatment for hyperhidrosis, such as anticholinergic drugs (e.g. glycopyrrolate), sedatives or tranquilizers, within the past 8 weeks.
3. Subjects who have undergone surgical excision of sweat glands or sympathectomy for hyperhidrosis.
4. Subjects with an underlying disorder, such as neurologic injury or disease affecting the autonomic system, vascular disorders and metabolic disorders (e.g. hyperthyroidism, diabetes mellitus) that can produce hyperhidrosis
5. Subjects with a history of coronary artery disease.
6. Subjects with a history of poor compliance or psychosis
7. Subjects taking SSRIs, SNRIs, TCAs, or MAOIs
8. Subjects with known hypersensitivity to methylene blue
9. Subjects with cardiac pacemaker or any other electrically powered implantable device.
10. Subjects not proficient in the English language.
11. Subject not in appropriate physical health to ride a stationary bicycle to the point of eliciting sweat.
12. Known allergy to iodine or potato starch.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Measurement of changes in sweat production using gravimetric method | Measured at multiple time points, last at 6 months
  Compare treated side to control side

CONTACTS AND LOCATIONS:
Overall Officials: R Rox Anderson, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital - Wellman Center for Photomedicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided